CLINICAL TRIAL: NCT00002085
Title: A Study to Evaluate the Safety and Efficacy of Azithromycin in Individual Patients With Serious Nontuberculous Mycobacterial Disease Who Are Failing or Intolerant of Other Available Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 058D; 066-169
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections; Tuberculosis, Mycobacterium Infection
Keywords: Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Azithromycin; Mycobacterium Infections, Atypical
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Tuberculosis; Acquired Immunodeficiency Syndrome; Mycobacterium Infections, Nontuberculous | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate the efficacy and safety of azithromycin given chronically for the treatment of serious nontuberculous mycobacterial infection in patients failing or intolerant of other available therapy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Other antimicrobial drugs as long as documented on Case Report Form.

Patients must have:

* Serious nontuberculous mycobacterial infection.
* Approval of eligibility from Pfizer Clinical Monitor. Patients below the legal age of consent must have consent of parent or guardian.

NOTE:

* Pregnant women, women of childbearing potential, and children will not be specifically excluded from participation. However, patients and physicians should be aware that the safety of azithromycin during pregnancy and in long-term use in children and adults has not been established. The risks and benefits of azithromycin use in these patients will be considered in consultation with the physician and the Pfizer Clinical Monitor.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Disseminated Mycobacterium avium complex (MAC) who are eligible for treatment with azithromycin under protocol 066-162.
* Known hypersensitivity or intolerance to macrolide antibiotics.

Patients with the following prior conditions are excluded:

History of hypersensitivity or intolerance to azithromycin.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pfizer Central Research, Groton, Connecticut
  - Natl Cancer Institute / Metabolism Branch, Bethesda, Maryland